CLINICAL TRIAL: NCT02752113
Title: ELMI - Prospective, Randomized, Controlled, Parallel-arm Study to Assess the Effects of the Combined Therapy of Empagliflozin and Linagliptin Compared to Metformin and Insulin Glargine on Renal and Vascular Changes in Type 2 Diabetes
Brief Title: Effects of Empagliflozin + Linagliptin vs Metformin + Insulin Glargine on Renal and Vascular Changes in Type 2 Diabetes
Acronym: ELMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPPMed-2016-01-ELMI; 2016-000242-57 (EudraCT Number)
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes mellitus type 2; Metformin; Micro- and macrocirculation; HbA1c >= 7%
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Linagliptin; Metformin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empagliflozin and Linagliptin (Active Comparator): After the 4 weeks run-in phase (stable metformin medication), patients will be consecutively randomized (1:1) to empagliflozin 10 mg and linagliptin 5 mg orally once daily. After 14 days empagliflozin will be up-titrated to 25 mg (once daily), if fasting blood glucose is ≥ 100 mg /dl and no hypoglycemic symptoms are recognized.
  Interventions: Drug: Empagliflozin and Linagliptin
- Metformin and Insulin sc (Active Comparator): Metformin p.o. and insulin sc After the 4 weeks run-in phase (stable metformin medication), patients will maintain on their metformin dosage (850 or 1000 mg orally twice daily) and insulin glargine (Lantus™) once daily subcutaneous will be added. Initially 2 - 4 U Lantus™ daily (depending on body weight) will be given, and adjusted every third day (telephone counseling) by adding 2 U if fasting blood glucose is not ≤ 125 mg/dl (16). After a stable dosage (i.e. no change of dosage for 1 week) has been reached, adjustments regarding an increment of Lantus™ will be based on confirmed fasting blood glucose of ≥ 126 mg/dl (on at least two consecutive day).
  Interventions: Drug: Metformin and Insulin sc

INTERVENTIONS:
Drug: Empagliflozin and Linagliptin — Empagliflozin and Linagliptin
  Other Names: Jardiance, Trajenta
  Arms: Empagliflozin and Linagliptin
Drug: Metformin and Insulin sc — Metformin and Insulin sc
  Other Names: Siofor, Lantus
  Arms: Metformin and Insulin sc

SUMMARY:
Diabetes mellitus is a wide-spread disease accompanied by strongly increased morbidity and mortality due to micro- and macrovascular complications. However, in studies with patients suffering from diabetes mellitus type 2 (DM 2), early changes and impairments in large and small blood vessels as well as organ damage (e. g. to the kidneys) have been only insufficiently investigated (1). The newest substance class in oral antidiabetics, i. e. SGLT-2-inhibitors (such as empagliflozin) cause an increased renal excretion of glucose. In addition, the concurrent increased sodium excretion brings about an improvement of vascular function and thus a decrease in blood pressure. In the EMP-REG-OUTCOME study (2), the cardiovascular mortality rate was significantly lower in the empagliflozin group (3.7% versus 5.9%; 38% relative RR) compared to placebo.For another new substance class, the dipeptidylpeptidase-4-inhibitors, a number of pleiotropic effects have been described (3). In one of our recently conducted trials, we could demonstrate a positive effect of linagliptin on renal an inflammatory parameters compared to placebo (4). Thus, the combination of both substance classes with regard to positive effects on micro- and macrocirculation, even though not sufficiently proven as yet, suggests itself. The therapy with metformin and long-acting insulin (BOT), as well as a twofold oral medication is possible according to the recommendations of the "Deutsche Diabetes Gesellschaft (DDG)" and the positional paper of the "American Diabetes Association (ADA)". Accordingly, the aim of the present paper is the analysis of the effects of a combined therapy with empagliflozin plus linagliptin compared to metformin plus insulin glargine on renal and vascular changes in type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus, considered at the beginning as a metabolic disorder, mutates into a predominantly vascular disease, once its duration extends over several years or/and when additional cardiovascular (CV) risk factors coexist, in particular arterial hypertension. As a consequence, treatment of type 2 diabetes should focus not only on metabolic control but also on improving the vascular structure and function in the micro- and macrocirculation (1). Glomerular hyperfiltration and hyperperfusion pointing to altered intraglomerular hemodynamics, e.g. reduced preglomerular (i.e. resistance of the afferent arteriole [Ra]) resistance and increased postglomerular (i.e. resistance of the efferent arteriole [Re]) resistance (resulting in an increased intraglomerular pressure [Pglom]) are considered to be pivotal hemodynamic hallmarks of renal impairment in early diabetes (2). Endothelium dysfunction is a key pathogenetic process leading to increased leakage of albumin through the glomerular barrier and represents a pivotal determinant of glomerular filtration rate (GFR) (3; 4). Poor glycemic control is related to hyperperfusion and increased basal nitric oxide (NO) activity secondary to increased oxidative stress that leads to impaired endothelial function in early diabetes (5). Indeed, endothelial function increased after reducing oxidative stress as evidenced by the results with the infusion of vitamin C (6). The assessment of pulse wave velocity (PWV), pulse wave analysis (PWA), central (aortic) systolic pressure and pulse pressure, forward and backward wave amplitude are tools to detect early vascular changes related to a faster wave reflection in the arterial tree and are considered valid intermediate (surrogate) endpoints of vascular damage (7; 8). These parameters are only infrequently measured in studies with type 2 diabetes (9), mainly due to lack of expertise required to assess these vascular and renal markers, and lack of awareness that vascular changes are the key prognostic factor in type 2 diabetes. Empagliflozin is a novel selective inhibitor of the sodium-glucose cotransporter 2 (SGLT-2) that has been shown to improve glycemic control after 12, and 24 weeks as well as after 1 year (10). Empagliflozin produced dose dependent increases in glucosuria and clinically meaningful changes of glycemic parameters in type 2 diabetes (e.g. Glycosylated Hemoglobin [HbA1c]), in addition to weight loss and blood pressure reduction. In parallel to glucosuria, sodium is excreted in the urine and loss of sodium leads to a less reactive contraction of the small arteries in response to sympathetic activity, angiotensin II and catecholamines. The reduction in blood pressure might be related to weight loss and loss of intravascular volume and sodium content as well as to improved vascular function. In the EMPA-REG-OUTCOME trial (11) the empagliflozin group had significantly lower rates of death from CV causes (3.7%, vs. 5.9% in the placebo group; 38% relative risk reduction), hospitalization for heart failure (2.7% and 4.1%, respectively; 35% relative risk reduction), and death from any cause (5.7% and 8.3%, respectively; 32% relative risk reduction). These beneficial effects on hard outcome parameters might be related to the effects of empagliflozin described above. Furthermore, among patients receiving empagliflozin, there was admittedly an increased rate of genital infection but no increased incidence in other adverse events or any other safety parameter was observed. Dipeptidyl peptidase-4 (DPP-4) inhibitors, the other new drug class of antidiabetic agents, are also attractive agents to treat type 2 diabetes. So far, the predominant focus was on its antidiabetic efficacy, but several pleiotropic effects of DPP-4 inhibitors have been described (12). Indeed, we observed beneficial renal effects with linagliptin, e.g. preserved preglomerular resistance and NO activity in the renal vascular bed, compared to placebo, as well as reduced inflammatory markers (13). Thus, to combine empagliflozin with linagliptin is obvious and the antiglycemic potency and safety have been and still are examined in a large phase 3 program (14). Moreover, due to the pleiotropic effects of these 2 compounds (described above), synergistic beneficial effects on the micro- and macrocirculation (vascular and renal effects) can be expected (though not yet proven) and may explain to great extent the observed beneficial effects of empagliflozin on CV death and total mortality (11). According to the guidelines the combination of insulin and metformin is still, however, considered a valid and well established combination to control hyperglycemia. However, according to the update of the Position Statement of the American Diabetes Association (ADA) and European Association for the Study of Diabetes (EASD) advancing to dual oral combination, and even triple oral antiglycemic therapy is a recommended alternative (15). Hence, at least when metformin is contraindicated or not tolerated, the combination of DPP-4 inhibitors and SGLT-2 inhibitors may be a preferably choice. The goal of the current proposal is to prove the hypothesis that at similar levels of glycemic control the combination empagliflozin and linagliptin exert beneficial effects on the renal and vascular endothelium and on vascular surrogate endpoints in patients with type 2 diabetes as opposed to the combination of metformin and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, using already metformin (850 or 1000 mg twice daily) for at least 2 months prior to screening visit or type 2 diabetes switched to metformin at least 3 months prior to randomisation visit
* HbA1c ≥6.5 % if on antidiabetic montherapy or HbA1c ≥ 6.0 if on two antidiabetic drugs - Age of 18 - 75 years
* Male and female patients (females of child bearing potential must be using adequate contraceptive precautions)
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at screening visit
* Informed consent (§ 40 Abs. 1 Satz 3 Punkt 3 AMG) has to be given in written form.

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Use of insulin, glitazone, gliptin or SGLT-2 inhibitor within the past 2 months
* HbA1c > 10.5% if on antidiabetic monotherapy and > 9.5% if on two antidiabetic drugs
* Fasting plasma glucose > 240 mg/dl
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 6 months prior to study inclusion
* UACR ≥ 300 mg/g (early morning spot urine)
* Estimated GFR (eGFR) < 60 ml/min/1.73m²
* Uncontrolled arterial hypertension (blood pressure ≥ 180/110 mmHg)
* Congestive heart failure NYHA stage III and IV
* Severe disorders of the gastrointestinal tract or other diseases which interfere the pharmacodynamics and pharmacokinetics of study drugs
* Significant laboratory abnormalities such as serum Glutamate-Oxaloacetate-Transaminase (SGOT) or serum Glutamate-Pyruvate-Transaminase (SGPT) levels more than 3 x above the upper limit of normal range
* Drug or alcohol abuses
* Pregnant or breast-feeding patients
* Use of loop diuretics
* History of repetitive urogenital infection per year
* Body mass index > 40 kg/m²
* Triglyceride levels > 1000 mg/dl
* High density lipoprotein (HDL)-cholesterol levels < 25 mg/dl
* Any patient currently receiving chronic (>30 consecutive days) treatment with an oral corticosteroid
* Patients being treated for severe auto immune disease e.g. lupus
* Participation in another clinical study within 30 days prior to visit 1
* Individuals at risk for poor protocol or medication compliance
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Effect of empagliflozin plus linagliptin vs metformin plus insulin glargine on basal NO activity of renal vasculature (response of RPF (renal plasma flow) to L-NMMA (NG-monomethyl-L-arginine) infusion) | at baseline and after 3 months on empagliflozin plus linagliptin or metformin plus insulin glargine, respectively
  Poor glycemic control is related to hyperperfusion and increased basal nitric oxide (NO) activity secondary to increased oxidative stress that leads to impaired endothelial function in early diabetes.

SECONDARY OUTCOMES:
Changes in oxidative stress level of renal vasculature (response of RPF to vitamin C infusion) | at baseline and after 3 months on empagliflozin plus linagliptin or metformin plus insulin glargine, respectively
changes in intraglomerular resistances (Ra and Re) and Pglom | at baseline and after three months
changes in albuminuria (urinary albumin to creatinine ratio [UACR]), assessed in the 24-hour urine | at baseline and after three months

CONTACTS AND LOCATIONS:
Overall Officials: Roland Schmieder, Prof MD, Principal Investigator — Department of Nephrology and Hypertension, University of Erlangen-Nuremberg; Peter Bramlage, Prof MD, Study Chair — IPPMed
Locations (1):
- Clinical Research Center, Dept of Nephrology and Hypertenison, University of Erlangen/Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Striepe K, Jumar A, Ott C, Karg MV, Schneider MP, Kannenkeril D, Schmieder RE. Effects of the Selective Sodium-Glucose Cotransporter 2 Inhibitor Empagliflozin on Vascular Function and Central Hemodynamics in Patients With Type 2 Diabetes Mellitus. Circulation. 2017 Sep 19;136(12):1167-1169. doi: 10.1161/CIRCULATIONAHA.117.029529. No abstract available. PMID 28923906
- [Derived] Gunes-Altan M, Bosch A, Striepe K, Bramlage P, Schiffer M, Schmieder RE, Kannenkeril D. Is GFR decline induced by SGLT2 inhibitor of clinical importance? Cardiovasc Diabetol. 2024 May 29;23(1):184. doi: 10.1186/s12933-024-02223-0. PMID 38811998
- [Derived] Staef M, Ott C, Kannenkeril D, Striepe K, Schiffer M, Schmieder RE, Bosch A. Determinants of arterial stiffness in patients with type 2 diabetes mellitus: a cross sectional analysis. Sci Rep. 2023 Jun 2;13(1):8944. doi: 10.1038/s41598-023-35589-4. PMID 37268640
- [Derived] Ott C, Jung S, Korn M, Kannenkeril D, Bosch A, Kolwelter J, Striepe K, Bramlage P, Schiffer M, Schmieder RE. Renal hemodynamic effects differ between antidiabetic combination strategies: randomized controlled clinical trial comparing empagliflozin/linagliptin with metformin/insulin glargine. Cardiovasc Diabetol. 2021 Sep 4;20(1):178. doi: 10.1186/s12933-021-01358-8. PMID 34481498
- [Derived] Jung S, Bosch A, Kannenkeril D, Karg MV, Striepe K, Bramlage P, Ott C, Schmieder RE. Combination of empagliflozin and linagliptin improves blood pressure and vascular function in type 2 diabetes. Eur Heart J Cardiovasc Pharmacother. 2020 Nov 1;6(6):364-371. doi: 10.1093/ehjcvp/pvz078. PMID 31816038